CLINICAL TRIAL: NCT01922817
Title: A Dipeptidyl Peptidase 4 (DPP-4) Inhibitor in Type 1 Diabetes
Brief Title: DPP4inhibitors in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2012DM07
Record Dates: First submitted 2013-08-06; First posted 2013-08-14 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes; Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — saxagliptin

STUDY DESIGN:
Intervention Model Description: crossover trial between Saxaglipin and Placebo with 2 week washout in between
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Active Comparator): 5mg once daily in addition to insulin therapy
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator): Crossover Placebo once daily
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — 5mg saxagliptin

SUMMARY:
A small, pilot, randomised, cross over trial that investigates the potential for DPPIVi therapy to reduce insulin requirements in type 1 diabetes was studied. We investigated whether this drug reduces daily insulin doses, leads to weight reduction, reduces blood glucose fluctuation and improves glucose control. Through reduction of blood glucose variability, we want investigated, whether it has the capability of improving the magnitude of epinephrine responses at 2.5mmol/L by performing a hyperinsulinaemic, hypoglycaemia clamp study after each arm. A successful outcome would then lead to an application for funds for a larger, multicentre intervention study. The benefits of this therapeutic advance are clear and this has the potential to make a dramatic improvement to the lives of people with type 1 diabetes in our community.

DETAILED DESCRIPTION:
Ninety years ago the discovery of insulin and its development as a drug revolutionized the management of type 1 diabetes, which until that point had almost inevitably proven fatal. However, very rapidly it was recognized that like all "wonder" drugs there were problems with insulin. Elliot Joslin, one of the pioneers of diabetes therapy described insulin as "…a potent preparation alike for evil and for good"(1922). There are two major reasons for this. Firstly, in non-diabetic individuals insulin produced by the pancreas acts directly on the liver, the major organ for regulating blood glucose levels. In contrast, people with type 1 diabetes inject insulin under the skin, and this is then absorbed into the circulation and much of it is degraded (~50%) before it gets to the liver. This means that in order to act effectively in the liver a type 1 diabetic needs to inject at least double the amount of insulin. Many studies have now shown that high insulin levels lead to weight gain, accelerated blood vessel disease (atherosclerosis) and a higher risk of suffering low blood glucose (hypoglycaemia). A second major problem is that individuals with type 1 show high levels of the hormone, glucagon. Glucagon is also produced in the pancreas and is normally regulated by pancreatic insulin, so the loss of this effect in people with type 1 diabetes means they run high glucagon levels. This has been shown to increase blood glucose, particularly after a meal. It is because of this that the diabetes community has called for novel therapies that can reduce high insulin levels and high glucagon levels. A new class of drugs called dipeptidylpeptidase IV inhibitors (DPPIVi) are currently used to treat people with type 2 diabetes. DPPIV inhibition increases endogenous levels of glucagon like peptide-1 (GLP-1). These drugs have a number of actions but the most relevant to this application is that they directly suppress glucagon, induce satiety (i.e. reduce hunger and leads to a reduction in body weight) and indirectly reduce the need for high dose insulin injections. This makes them an ideal candidate drug as an insulin sparing or adjunct therapy in type 1 diabetes, but there is very limited data to date for this use.

ELIGIBILITY:
Inclusion criteria;

* Type 1 diabetes over 5 years duration
* HbA1c less than 10%
* Age 18 and over
* Current use of intensive insulin therapy (injections or pump)
* BMI 19-35
* Ability to give written informed consent to participate in the study

Exclusion criteria;

* Previous history of pancreatic disease/cancer
* Significant renal disease estimated glomerular filtration rate (eGFR) less than 50
* Significant microvascular disease
* Personal/family history of Medullary thyroid cancer
* Personal/family history of multiple endocrine neoplasia (MEN) Type 2
* Moderate/Severe hepatic impairment
* Pregnancy or breast feeding
* History of epilepsy/hypoglycaemia induced seizure
* Those on any other hypoglycaemia drug apart from insulin for their diabetes.
* Currently on CYP3A4 inducers like carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampicin
* Currently on CYP3A4 inhibitors like ketoconazole, diltiazem
* Less than 30 days since participation in another drug trial or longer depending on the drug half life.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Magnitude of epinephrine release at 2.5mmol/L | During hyperinsulinaemic hypoglycaemia clamp

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical research centre, Ninewells Hospital and Medical School, Dundee, United Kingdom

REFERENCES:
- [Background] George PS, McCrimmon RJ. Saxagliptin co-therapy in C-peptide negative Type 1 diabetes does not improve counter-regulatory responses to hypoglycaemia. Diabet Med. 2016 Sep;33(9):1283-90. doi: 10.1111/dme.13046. Epub 2015 Dec 28. PMID 26642301